CLINICAL TRIAL: NCT06166550
Title: Improving Psychological Wellbeing Through Stress Reduction Among Parents Having Children With Neurodevelopmental Disorders: A Multi-pronged Intervention in Bangladesh
Brief Title: Improving Psychological Wellbeing by Stress Reduction Among Parents Having Children With Neurodevelopmental Disorders
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Bangabandhu Sheikh Mujib Medical University, Dhaka, Bangladesh (Other)
Collaborators: Centre for Injury Prevention and Research Bangladesh (Other); University of Dhaka, Bangladesh (Other); Directorate General of Health Services, Ministry of Health and Family Welfare, Bangladesh (Unknown)
Responsible Party: Principal Investigator, Md Atiqul Haque, Dean and Chairman, Bangabandhu Sheikh Mujib Medical University, Dhaka, Bangladesh
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: BSMMU/2022/10733
Record Dates: First submitted 2023-10-10; First posted 2023-12-12 (Actual); Last update posted 2025-08-22 (Actual); Status verified 2025-08

CONDITIONS: Mental Health Issue
Keywords: Psychological wellbeing; Neurodevelopmental Disorder; Parental Stress; Emotional Intelligence
MeSH Terms: conditions — Neurodevelopmental Disorders | interventions — Medical Records

STUDY DESIGN:
Intervention Model Description: The intervention is based on Emotional Intelligence. A training session will be given in-person; a diary and a mobile app will be given to practice emotional intelligence at home.
Who Masked: Outcomes Assessor
Masking Description: The arms will be labelled as group A and group B. The statisticians will be blind about the labelling. Thus, the masking will be ensured.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention (Experimental): Parents of children suffering from neurodevelopmental disorders will be the participants. They will get in-person training on emotional intelligence and access to a mobile app and a personal diary aimed at enhancing their psychological wellbeing.
  Interventions: Behavioral: Parent's Emotional Intelligence Network; Device: Mobile App; Device: Diary
- Control (No Intervention): This group will be in wait-list, get no intervention at the initial phase. They will get the intervention after the intervention period and the endline survey is over.

INTERVENTIONS:
Behavioral: Parent's Emotional Intelligence Network — A two-day in-person training session will be arranged for the participating parents at least one week apart. The psychologists will conduct the training session on emotional intelligence. A training of the trainer manual will be developed to train the psychologists. The training session will include a power point presentation and certain group and individual activities to practice emotional intelligence. The participants will also be given a diary and a mobile app in order to practice emotional intelligence at home.
  Arms: Intervention
Device: Mobile App — A mobile app (MonKotha) has been developed along with user manual. It contains different videos, audios, and texts related to emotional intelligence. It also provides a communication platform where users can communicate through texts and upload documents.
  Other Names: MonKotha - A parents' emotional intelligence network
  Arms: Intervention
Device: Diary — A diary (Onuvutir Diary) is also developed that contain different practice materials regarding emotional intelligence. It is a personal diary given to the participants to take to home.
  Other Names: Onuvutir Diary
  Arms: Intervention

SUMMARY:
This project addresses the mental health challenges faced by parents caring for children with Neurodevelopmental Disorders (NDDs) in Bangladesh. These parents often experience high levels of stress, anxiety, and depression, impacting family dynamics and the child's development. The project aims to design, implement, and assess an intervention to reduce parenting stress and enhance parental well-being. This intervention focuses on emotional intelligence and will be delivered through in-person training and a mobile app. The study will use a cluster randomized controlled trial methodology, targeting parents of children diagnosed with NDDs.

The study will be conducted in Child Development Centers in public medical college hospitals across Bangladesh. It will assess changes in parental stress, mental well-being, and emotional intelligence. Data collection will occur from January 2024 to June 2025.

The project aims to recruit 480 parents from eight Child Development Centers, ensuring ethical considerations, data integrity, and participant privacy. The findings will be shared through national dissemination seminars, policy briefs, reports, and journal publications.

DETAILED DESCRIPTION:
Background and Rationale:

Neurodevelopmental disorders (NDDs) are a global public health concern, often causing parents to grapple with increased stress, anxiety, and reduced well-being. This compromised mental health among caregivers persists throughout a child's development, straining family dynamics and making effective parenting more challenging. Research underscores the importance of addressing caregiver's well-being, as it indirectly impacts the child's health and development.

In Bangladesh, where social stigma and limited support exacerbate the challenges, there is a lack of research on stress management to improve parental well-being. Empirical studies are essential to enhance the psychological health of caregivers of children with NDDs in Bangladesh and promote long-term caregiving abilities.

Objectives:

The project aims to develop an evidence-based intervention to reduce parenting stress and enhance the mental health of parents with children with neurodevelopmental disorders. This intervention will be implemented in healthcare and community settings and evaluated through process and outcome measures, including changes in parenting stress.

Trial design:

The trial will adopt a parallel design and employ a cluster randomized controlled trial (CRCT) methodology.

Methods:

Study settings:

The study is centered around the Institute of Paediatric Neurology and Autism (IPNA) and Child Development Centers or Shishu Bikash Kendra (SBKs) in Bangladesh's eight administrative divisions. IPNA at BSMMU provides care, education, and training, impacting national mental health policy. Additionally, fifteen government medical college hospitals operate SBKs as outdoor services. These centers offer specialized care for children with NDDs through a multidisciplinary team.

Eligibility criteria:

Parents aged 18 to 50 years with children having neurodevelopmental disorders (e.g., Autism, Cerebral Palsy, Intellectual disorders, ADHD, and Down Syndrome) diagnosed at the SBKs are eligible. Exclusions include parents of children with sensory impairments, oxygen-dependent chronic lung disorders, or requiring initial pharmacological care. An implementation guide will be created, facilitators trained in emotional intelligence, and community mobilizers trained for SBK-based campaigns to ensure smooth intervention implementation.

Intervention:

Investigators will develop an intervention module and a mobile app/software for parents of children with NDDs. The intervention will focus on enhancing emotional intelligence and stress reduction, with two interactive sessions covering emotional awareness, regulation, empathy, and interpersonal skills. Two groups will be involved: Group A (Training, diary & app users), and Group B (Control). Group A will receive in-person training and access to the app, and Group B will be in wait-list control group. The wait-list control group will receive the intervention after the intervention period is over. The aim is to improve emotional intelligence to handle life's stress. Morning and evening sessions will be available for working parents, and those needing pharmacological management will be referred to relevant department. The mobile app/software and the diary will support parents in improving emotional intelligence skills, benefiting family well-being and the child with special needs.

Outcomes:

This study's aim to assess the intervention's effectiveness and feasibility in Bangladesh's Child Development Centers and among the targeted parents. Parenting stress and psychological well-being will be evaluated. Secondary outcomes include mental health, emotional intelligence, parenting self-efficacy, perceived social support, parenting satisfaction, and marital satisfaction during the same period.

Sample Size and recruitment process:

Investigators used a sample size calculator to determine the sample size. The average cluster size will be 60 and cluster number will be 8. Adjusted for clusters, the maximum sample size is 480 parents. Eight SBKs, one per administrative division, will be randomly assigned to intervention and control groups in a 1:1 ratio. Lists of recently diagnosed children will be obtained. Investigators will invite both parents and continue recruiting until reaching the required sample size.

Methods:

Data Collection methods and data management:

Data collection steps involve contacting prospective parents to participate. Baseline data collection occurs at selected SBKs with self-administered questionnaires on parenting style, stress, and mental health. Groups A will receive the intervention, while Group B serves as the control. Follow-up evaluations at 12 weeks will measure stress and well-being. After follow-up data collection is over, Group B will receive the intervention.

Statistical methods:

Principles of analysis: The population for the primary outcome analysis will consist of all recruited parents who received two sessions of intervention and for whom both baseline and post intervention follow-up data will be available. If a participant moves to the catchment area of another SBK after baseline measure is collected (i.e., crossover from intervention to control, or vice versa), the instances will be documented, and removed from the trial. As the final population in the primary analysis will exclude the participants who will be lost to follow-up (i.e., for whom follow-up data is not available), a sensitivity analysis will be performed to account for all randomized participants.

Descriptive analysis: Socio-demographic data of the participants e.g., gender, occupation, education status, family history of neurodevelopmental disorders, etc. will be obtained. All categorical variables will be summarized in frequency and percentages, and continuous variables in mean and standard deviation. To estimate the association of these characteristics with parenting stress and psychological wellbeing, t-tests and chi-square tests will be done.

Inferential analysis: To estimate the efficacy of the intervention, before-after data will be analyzed, and paired t-test and McNemar's chi-square tests will be done in this regard. A comparison will also be made between the intervention and the control data, both at pre- and post- intervention level. Difference-in-difference analysis will be done to estimate the intervention effects among participants by age groups, sex, socio-economic status, etc.

Association analysis: Binary regression analysis will be done to estimate the association between socio-demographic variables with changes in the outcome variables, change in parenting stress and psychological wellbeing.

Data monitoring:

The Data Monitoring Committee (DMC) plays a vital role in ensuring the study's integrity and security. Comprising impartial specialists in mental health, neurodevelopmental disorders, and research ethics, DMC will independently monitor the study. DMC's main responsibility is to safeguard participants' rights and well-being by examining data, tracking study progress, and assessing risks or adverse outcomes related to the intervention. The DMC also ensures research techniques and analyses are appropriate and objective, maintaining scientific rigor. Ultimately, DMC will provide essential oversight, enhancing credibility, and upholding ethical standards while advancing knowledge in neurodevelopmental disorders and parental well-being.

Ethics and dissemination:

An informed consent will be sought from each participant prior to the collection of data, detailing the study's objectives, procedures, advantages, risks, and the identity of the lead investigator. This research protocol has received approval from the Institutional Review Board at BSMMU. Participants will be given unique ID numbers, and all information will be encrypted and kept confidential to preserve privacy, anonymity, and secrecy. The information gathered will only be utilized for study.

Confidentiality:

Local-level problems including non-cooperation and non-response are anticipated hurdles and barriers. These issues will be handled by rapport-building, sensitivity, and choosing the right responders. Respondents will be guaranteed of the privacy of data while confidentiality will be upheld. Following governmental directives, general contextual elements will be managed. The management of capacity issues and team dropout will involve ongoing observation, communication, and additional training.

Dissemination policy:

In this project, investigators are committed to share research findings widely for maximum impact. The dissemination strategy includes publishing in open-access academic journals, creating plain language summaries for accessibility, participating in conferences to engage with experts and practitioners, conducting community workshops, developing policy briefs for government agencies, collaborating with NGOs, and responsibly sharing de-identified data with fellow researchers. The goal is to reach a diverse audience, including parents, healthcare professionals, policymakers, and researchers, to enhance the well-being of parents and children with neurodevelopmental disorders in Bangladesh and beyond.

ELIGIBILITY:
Inclusion Criteria:

* Parents of any age having children with neurodevelopmental disorders i.e. Autism Spectrum Disorders, Cerebral Palsy, Intellectual disorders, attention deficit hyperactivity disorders, and Down Syndrome.
* Parents of children whose diagnosis were made within one year (to avoid the time-effect on stress and mental health).
* Parents' age limit will be 18-50 years

Exclusion Criteria:

* Parents having children with serious sensory impairments (e.g., deafness and blindness) and oxygen dependence due to chronic lung diseases.
* Parents who need pharmacological management at initial assessment.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 480 (Actual)
Dates: Start 2024-01-27 (Actual); Primary Completion 2025-06-30 (Actual); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Psychological well-being | 12 weeks after completion of the intervention
  Psychological well-being: The WHO-5 Well-Being Index will assess participants' subjective well-being before and after the intervention. Raw scores range from 0 to 25, with higher scores indicating better well-being.
Parenting stress | 12 weeks after completion of two-day intervention
  Parenting stress will be assessed by Parental Stress Scale, a 18-item Likert scale.
  Parental stress scores range from 18 to 90, with lower scores indicating lower levels of parental stress.
Mental Health | 12 weeks after the intervention.
  Mental health will be assessed using Depression, Anxiety, and Stress scale (DASS-9), a validated screening tool measuring depression, anxiety, and stress. Raw score ranges from 0 to 27, with higher score indicating more depression, anxiety, and stress.

SECONDARY OUTCOMES:
Emotional intelligence | 12 weeks after completion of the intervention
  Parent's emotional intelligence will be assessed by Trait Emotional Intelligence Questionnaire-Short Form (TEIQue-SF). The response scale is a 7-point Likert scale, ranging from 1 to 7. Greater scores represent better emotional intelligence.
Parenting Self-Efficacy | 12 weeks after completion of two-day intervention
  Parenting Self-Efficacy will be measured by parenting Self-Efficacy scale. Scores range from 5 to 25, with higher scores indicating greater self-efficacy.
Parenting satisfaction | 12 weeks after the completion of the intervention
  The Kansas Parental Satisfaction Scale will assess parenting satisfaction using a 7-point scale from extremely dissatisfied to extremely satisfied. Scores will range from 3 to 21, where greater scores represent better parental satisfaction.
Marital satisfaction | 12 weeks after the intervention
  The Kansas Marital Satisfaction Scale is designed to assess satisfaction in relationships among married couples. Scores will range from 3 to 21, where greater scores represent better marital satisfaction.
Fidelity | Perioperative.
  Fidelity will be assessed by recording all the intervention sessions. The fidelity scale, developed for this study, will be used to rate the components of the intervention on a rating scale (0 = Not Implemented, 1 = Poor Implementation, 2 = Partial/Moderate Implementation, and 3 = Fully Implemented as Intended). The following fidelity outcomes will be measured: Intervention-specific fidelity rate (e.g., Adherence to manual, use of materials, supervision and feedback, cultural and contextual fit), Adherence rate to protocol, Exposure, Quality of intervention delivery, and Participant's responsiveness.

CONTACTS AND LOCATIONS:
Overall Officials: Salim M Chowdhuri, PhD, Study Director — Center for Injury Prevention and Research Bangladesh
Locations (1):
- Bangabandhu Sheikh Mujib Medical University, Dhaka, Bangladesh

IPD SHARING:
Plan to Share IPD: Yes
Access to trial IPD can be requested by qualified researchers engaging in independent scientific research, and will be provided following review and approval of a research proposal and Statistical Analysis Plan (SAP) and execution of a Data Sharing Agreement (DSA).
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: The data will be made available after six months of the study completion and will be made accessible for up to 24 months.
Access Criteria: Access to trial IPD can be requested by qualified researchers engaging in independent scientific research, and will be provided following review and approval of a research proposal and Statistical Analysis Plan (SAP) and execution of a Data Sharing Agreement (DSA).

REFERENCES:
- [Derived] Salwa M, Chowdhury SM, Rois R, Uddin MK, Akhter S, Nahar K, Mullick AR, Mannan M, Kundu GK, Fatema K, Maruf Haque Khan M, Haque MA. Leveraging emotional intelligence to alleviate mental health: protocol of a cluster randomised controlled trial among parents of children with neurodevelopmental disorders in Bangladesh. BMJ Open. 2025 Sep 30;15(9):e105688. doi: 10.1136/bmjopen-2025-105688. PMID 41027705